CLINICAL TRIAL: NCT00408278
Title: Treatment of Newly Diagnosed Patients With Acute Promyelocytic Leukemia (PETHEMA LPA 2005): Remission Induction With ATRA + Idarubicin. Risk-adapted Consolidation With ATRA and Anthracycline-based Chemotherapy (Idarubicin/Mitoxantrone) With Addition of Ara-C for High-risk Patients. Maintenance Therapy With ATRA + Low Dose Chemotherapy (Methotrexate + Mercaptopurine).
Brief Title: Treatment of Newly Diagnosed Patients With Acute Promyelocytic Leukemia (PETHEMA LPA 2005)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPA 2005
Record Dates: First submitted 2006-12-05; First posted 2006-12-06 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: Acute Promyelocytic Leukemia
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Idarubicin; Mitoxantrone; Cytarabine

INTERVENTIONS:
Drug: ATRA — 45 mg/m2 day until CR Consolidation: 3 cycles (45 mg/m2 days 1-15) Maintenance:15 days every 3 months
Drug: Idarubicina — Induction: 12 mg/m2 days 2, 4, 6 and 8 Consolidation: 5 mg/m2 days 1-4 in cycle 1 and 12 mg/m2 day 1 in cycle 3.
Drug: Mitoxantrone — Consolidation: Mitoxantrone 10 mg/m2 days 1-3 in cycle 2
Drug: ARA-C — In high risk patients, consolidation with ara-C in cycles 1 and 3.

SUMMARY:
Primary objectives

* To evaluate the efficacy and toxicity of a risk-adapted protocol that use idarubicin for induction and consolidation therapy in patients with APL.
* To evaluate the impact of mitoxantrone reduction on the event-free, disease-free, and overall survival, as well as on the duration of remission and cumulative incidence of relapse in low- and intermediate-risk patients with APL.
* To evaluate the impact of the addition of ara-C to idarubicin courses of consolidation for high-risk patients (administered as in the original GIMEMA protocols) on the event-free, disease-free, and overall survival, as well as on the duration of remission and cumulative incidence of relapse.
* To evaluate the toxicity of the induction, consolidation, and maintenance chemotherapy in the whole series and in each treatment group in patients with APL.

Secondary objectives

• To compare all outcomes with those achieved with the PETHEMA LPA99 protocol.

DETAILED DESCRIPTION:
Treatment of induction with the simultaneous administration of ATRA (45 mg/m2 day until the RC) and idarubicine (12 mg/m2 days 2, 4, 6 and 8), 3 monthly cycles of consolidation with ATRA (45 mg/m2 days 1-15) and idarubicine (5 mg/m2 days 1-4) in the cycle #1, mitoxantrone (10 mg/m2 days 1-3) in the cycle #2 and idarubicine (12 mg/m2 day 1) in the cycle #3. The consolidation was reinforced for the group of patients with intermediate risk by means of an increase of the idarubicine to 7 mg in the cycle #1 and to 2 days in the cycle #3. In the patients of high risk, the consolidation was reinforced with the addition of altar-c in the cycles #1 and #3. For the maintenance treatment, one will administer to intermittent ATRA (15 days every 3 months) and chemotherapy low doses with methotrexate and 6-mercaptopurina during two years

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 75 years.
* ECOG ≤ 3.
* Morphologic Diagnosis of LPA (FAB M3 or variant M3). Those cases without typical morphology but with PML-RARα reordering also must be including.
* Genetic Diagnosis: t (15; 17) demonstrated by cariotipo conventional, FISH, PML-RARα reordering detected by RT-PCR or a pattern microspeckled demonstrated with antibody anti-PML (positive PGM3). Obvious, it will be had the result of these tests once initiated the treatment on the basis of a suspicion diagnoses morphologic

Exclusion Criteria:

* Age >75 years (the treatment with this protocol can be considered individually)
* Absence of PML-Rare reordering.
* To have received previously some type of treatment for LPA, including chemotherapy or retinoides. The previous treatment with corticoids, hidroxiurea or leucoaféresis is not reason for exclusion.
* To have received chemotherapy or x-ray for the treatment of a disease vitiates previous.
* Associate Neoplasia.
* Serious psychiatric Disease.
* Seropositividad for VIH.
* Contraindication to receive intensive chemotherapy, specially antraciclinas.
* Sérica Creatinina ≥ 2,5 mg/dL (≥ 250 μmol/l).
* Bilirrubina, fosfatasa alkaline, or GOT > 3 times the normal limit
* Test of positive pregnancy.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2005-07; Primary Completion 2012-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy and toxicity of a risk-adapted protocol that use idarubicin for induction and consolidation therapy in patients with APL. | 1 year
To evaluate the impact of mitoxantrone reduction on the event-free, disease-free, and overall survival. | 1 year
To evaluate the impact of the addition of ara-C to idarubicin courses of consolidation for high-risk patients on the event-free, disease-free, and overall survival | 1 year
To evaluate the toxicity of the induction, consolidation, and maintenance chemotherapy in the whole series and in each treatment group in patients with APL. | 1 year

SECONDARY OUTCOMES:
To compare all outcomes with those achieved with the PETHEMA LPA99 protocol. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: San Miguel Miguel Angel, Dr, Study Chair — Hospital La Fe de Valencia; Vellenga Edo, Dr, Study Director — Stichting Hemato-Oncologie voor Volwassenen Nederland; Lowenberg Bob, Dr, Study Director — Stichting Hemato-Oncologie voor Volwassenen Nederland
Locations (42):
- PALG, Lodz, Poland
- Spain (40):
  - Hospital Juan Canalejo, A Coruña
  - Hospital General, Albacete
  - Hospital general, Alicante
  - Hospital germans Trias i Pujol, Badalona
  - Hospital Clinic, Barcelona
  - Hospital de Sant Pau, Barcelona
  - Institut Català d'Oncologái, Barcelona
  - Basurtuko Ospitalea, Bilbao
  - Hospital general, Castellon
  - Hospital de Fuenlabrada, Fuenlabrada
  - Hospital "Dr. Trueta", Girona
  - Hospital de Jerez de la Frontera, Jerez de la Frontera
  - Hospital Insular de las Palmas, Las Palmas de Gran Canaria
  - Complejo Hospitalario León, León
  - Complexo Hospitalario Xeral-Calde, Lugo
  - Hospital 12 de Octubre, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Reina Sofia, Madrid
  - Hospital San Pedro de Alcántara, Madrid
  - Hospital Severo Ochoa, Madrid
  - H. Carlos Haya, Málaga
  - H. Universitario Virgen de la Victoria, Málaga
  - Hospital Sta. Maria del Rosell, Murcia
  - Hospital Central de Asturias, Oviedo
  - Hospital Dr Negrín, Palma de Gran Canaria
  - Hospital de Navarra, Pamplona
  - Hospital de Montecelo, Pontevedra
  - Hospital Clínico Universitario, Salamanca
  - Hospital de Cruces, Santander
  - Hospital de Santiago de Compostela, Santiago de Compostela
  - H.U. Virgen del Rocio, Seville
  - Hospital Joan XXIII, Tarragona
  - Hospital Dr. Peset, Valencia
  - Hospital general, Valencia
  - Hospital La Fe, Valencia
  - Hospital Clínico de Valladolid, Valladolid
  - Hospital Txagorritxu, Vitoria-Gasteiz
  - Hospital Virgen de la Concha, Zamora
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- Hospital Maciel, Montevideo, Uruguay

REFERENCES:
- [Background] Tallman MS, Nabhan C, Feusner JH, Rowe JM. Acute promyelocytic leukemia: evolving therapeutic strategies. Blood. 2002 Feb 1;99(3):759-67. doi: 10.1182/blood.v99.3.759. PMID 11806975
- [Background] Ohno R, Asou N, Ohnishi K. Treatment of acute promyelocytic leukemia: strategy toward further increase of cure rate. Leukemia. 2003 Aug;17(8):1454-63. doi: 10.1038/sj.leu.2403031. PMID 12886231
- [Background] Sanz MA, Martin G, Lo Coco F. Choice of chemotherapy in induction, consolidation and maintenance in acute promyelocytic leukaemia. Best Pract Res Clin Haematol. 2003 Sep;16(3):433-51. doi: 10.1016/s1521-6926(03)00040-9. PMID 12935961
- [Background] Asou N, Adachi K, Tamura J, Kanamaru A, Kageyama S, Hiraoka A, Omoto E, Akiyama H, Tsubaki K, Saito K, Kuriyama K, Oh H, Kitano K, Miyawaki S, Takeyama K, Yamada O, Nishikawa K, Takahashi M, Matsuda S, Ohtake S, Suzushima H, Emi N, Ohno R. Analysis of prognostic factors in newly diagnosed acute promyelocytic leukemia treated with all-trans retinoic acid and chemotherapy. Japan Adult Leukemia Study Group. J Clin Oncol. 1998 Jan;16(1):78-85. doi: 10.1200/JCO.1998.16.1.78. PMID 9440726
- [Background] Burnett AK, Grimwade D, Solomon E, Wheatley K, Goldstone AH. Presenting white blood cell count and kinetics of molecular remission predict prognosis in acute promyelocytic leukemia treated with all-trans retinoic acid: result of the Randomized MRC Trial. Blood. 1999 Jun 15;93(12):4131-43. PMID 10361110
- [Background] Fenaux P, Chastang C, Chevret S, Sanz M, Dombret H, Archimbaud E, Fey M, Rayon C, Huguet F, Sotto JJ, Gardin C, Makhoul PC, Travade P, Solary E, Fegueux N, Bordessoule D, Miguel JS, Link H, Desablens B, Stamatoullas A, Deconinck E, Maloisel F, Castaigne S, Preudhomme C, Degos L. A randomized comparison of all transretinoic acid (ATRA) followed by chemotherapy and ATRA plus chemotherapy and the role of maintenance therapy in newly diagnosed acute promyelocytic leukemia. The European APL Group. Blood. 1999 Aug 15;94(4):1192-200. PMID 10438706
- [Background] Lengfelder E, Reichert A, Schoch C, Haase D, Haferlach T, Loffler H, Staib P, Heyll A, Seifarth W, Saussele S, Fonatsch C, Gassmann W, Ludwig WD, Hochhaus A, Beelen D, Aul C, Sauerland MC, Heinecke A, Hehlmann R, Wormann B, Hiddemann W, Buchner T. Double induction strategy including high dose cytarabine in combination with all-trans retinoic acid: effects in patients with newly diagnosed acute promyelocytic leukemia. German AML Cooperative Group. Leukemia. 2000 Aug;14(8):1362-70. doi: 10.1038/sj.leu.2401843. PMID 10942230
- [Background] Sanz MA, Lo Coco F, Martin G, Avvisati G, Rayon C, Barbui T, Diaz-Mediavilla J, Fioritoni G, Gonzalez JD, Liso V, Esteve J, Ferrara F, Bolufer P, Bernasconi C, Gonzalez M, Rodeghiero F, Colomer D, Petti MC, Ribera JM, Mandelli F. Definition of relapse risk and role of nonanthracycline drugs for consolidation in patients with acute promyelocytic leukemia: a joint study of the PETHEMA and GIMEMA cooperative groups. Blood. 2000 Aug 15;96(4):1247-53. PMID 10942364
- [Background] Sanz MA, Martin G, Gonzalez M, Leon A, Rayon C, Rivas C, Colomer D, Amutio E, Capote FJ, Milone GA, De La Serna J, Roman J, Barragan E, Bergua J, Escoda L, Parody R, Negri S, Calasanz MJ, Bolufer P; Programa de Estudio y Traitmiento de las Hemopatias Malignas. Risk-adapted treatment of acute promyelocytic leukemia with all-trans-retinoic acid and anthracycline monochemotherapy: a multicenter study by the PETHEMA group. Blood. 2004 Feb 15;103(4):1237-43. doi: 10.1182/blood-2003-07-2462. Epub 2003 Oct 23. PMID 14576047
- [Background] Grimwade D, Gorman P, Duprez E, Howe K, Langabeer S, Oliver F, Walker H, Culligan D, Waters J, Pomfret M, Goldstone A, Burnett A, Freemont P, Sheer D, Solomon E. Characterization of cryptic rearrangements and variant translocations in acute promyelocytic leukemia. Blood. 1997 Dec 15;90(12):4876-85. PMID 9389704
- [Background] van Dongen JJ, Macintyre EA, Gabert JA, Delabesse E, Rossi V, Saglio G, Gottardi E, Rambaldi A, Dotti G, Griesinger F, Parreira A, Gameiro P, Diaz MG, Malec M, Langerak AW, San Miguel JF, Biondi A. Standardized RT-PCR analysis of fusion gene transcripts from chromosome aberrations in acute leukemia for detection of minimal residual disease. Report of the BIOMED-1 Concerted Action: investigation of minimal residual disease in acute leukemia. Leukemia. 1999 Dec;13(12):1901-28. doi: 10.1038/sj.leu.2401592. PMID 10602411
- [Background] Falini B, Flenghi L, Fagioli M, Lo Coco F, Cordone I, Diverio D, Pasqualucci L, Biondi A, Riganelli D, Orleth A, Liso A, Martelli MF, Pelicci PG, Pileri S. Immunocytochemical diagnosis of acute promyelocytic leukemia (M3) with the monoclonal antibody PG-M3 (anti-PML). Blood. 1997 Nov 15;90(10):4046-53. PMID 9354674
- [Background] Gomis F, Sanz J, Sempere A, Plume G, Senent ML, Perez ML, Cervera J, Moscardo F, Bolufer P, Barragan E, Martin G, Sanz MA. Immunofluorescent analysis with the anti-PML monoclonal antibody PG-M3 for rapid and accurate genetic diagnosis of acute promyelocytic leukemia. Ann Hematol. 2004 Nov;83(11):687-90. doi: 10.1007/s00277-004-0902-7. Epub 2004 Jul 24. PMID 15278297
- [Derived] Martinez-Cuadron D, Montesinos P, Vellenga E, Bernal T, Salamero O, Holowiecka A, Brunet S, Gil C, Benavente C, Ribera JM, Perez-Encinas M, De la Serna J, Esteve J, Rubio V, Gonzalez-Campos J, Escoda L, Amutio ME, Arnan M, Arias J, Negri S, Lowenberg B, Sanz MA. Long-term outcome of older patients with newly diagnosed de novo acute promyelocytic leukemia treated with ATRA plus anthracycline-based therapy. Leukemia. 2018 Jan;32(1):21-29. doi: 10.1038/leu.2017.178. Epub 2017 Jun 6. PMID 28584252
- [Derived] Sanz MA, Montesinos P, Kim HT, Ruiz-Arguelles GJ, Undurraga MS, Uriarte MR, Martinez L, Jacomo RH, Gutierrez-Aguirre H, Melo RA, Bittencourt R, Pasquini R, Pagnano K, Fagundes EM, Vellenga E, Holowiecka A, Gonzalez-Huerta AJ, Fernandez P, De la Serna J, Brunet S, De Lisa E, Gonzalez-Campos J, Ribera JM, Krsnik I, Ganser A, Berliner N, Ribeiro RC, Lo-Coco F, Lowenberg B, Rego EM; IC-APL and PETHEMA and HOVON Groups. All-trans retinoic acid with daunorubicin or idarubicin for risk-adapted treatment of acute promyelocytic leukaemia: a matched-pair analysis of the PETHEMA LPA-2005 and IC-APL studies. Ann Hematol. 2015 Aug;94(8):1347-56. doi: 10.1007/s00277-015-2393-0. Epub 2015 May 15. PMID 25975975
- [Derived] Montesinos P, Rayon C, Vellenga E, Brunet S, Gonzalez J, Gonzalez M, Holowiecka A, Esteve J, Bergua J, Gonzalez JD, Rivas C, Tormo M, Rubio V, Bueno J, Manso F, Milone G, de la Serna J, Perez I, Perez-Encinas M, Krsnik I, Ribera JM, Escoda L, Lowenberg B, Sanz MA; PETHEMA; HOVON Groups. Clinical significance of CD56 expression in patients with acute promyelocytic leukemia treated with all-trans retinoic acid and anthracycline-based regimens. Blood. 2011 Feb 10;117(6):1799-805. doi: 10.1182/blood-2010-04-277434. Epub 2010 Dec 8. PMID 21148082
- [Derived] Sanz MA, Montesinos P, Rayon C, Holowiecka A, de la Serna J, Milone G, de Lisa E, Brunet S, Rubio V, Ribera JM, Rivas C, Krsnik I, Bergua J, Gonzalez J, Diaz-Mediavilla J, Rojas R, Manso F, Ossenkoppele G, Gonzalez JD, Lowenberg B; PETHEMA and HOVON Groups. Risk-adapted treatment of acute promyelocytic leukemia based on all-trans retinoic acid and anthracycline with addition of cytarabine in consolidation therapy for high-risk patients: further improvements in treatment outcome. Blood. 2010 Jun 24;115(25):5137-46. doi: 10.1182/blood-2010-01-266007. Epub 2010 Apr 14. PMID 20393132
- See also: Spanish association of Haematology — http://www.aehh.org
- See also: Hovon Data Center — http://www.hovon.nl